CLINICAL TRIAL: NCT06317298
Title: Efficacy and Safety of Fruquintinib in Combination With Everolimus as Second Line Therapy of ccRCC Patients Progressed Post Immunotherapy and Tyrosine Kinase Inhibitors Therapy: a Prospective, Single Arm, Phase II Clinical Trial
Brief Title: Fruquintinib Plus Everolimus as 2nd Line Therapy of ccRCC Patients Progressed Post IO and TKI Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-013-CH01 IIT-RCC
Record Dates: First submitted 2023-12-05; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Renal Cell Carcinoma, Clear Cell, Somatic
Keywords: fruquintinib; everolimus
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — HMPL-013; Everolimus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fruquintinib(3mg) plus Everolimus (Experimental): Fruquintinib 3mg Qd 21 days on 7 days off; Everolimus 5mg Qd; 28 day cycle until disease progression or intolerable adverse events
  Interventions: Drug: Fruquintinib and Everolimus
- Fruquintinib(4mg) plus Everolimus (Experimental): Fruquintinib 4mg Qd 21 days on 7 days off; Everolimus 5mg Qd; 28 day cycle until disease progression or intolerable adverse events
  Interventions: Drug: Fruquintinib and Everolimus
- Fruquintinib(5mg) plus Everolimus (Experimental): Fruquintinib 5mg Qd 21 days on 7 days off; Everolimus 5mg Qd; 28 day cycle until disease progression or intolerable adverse events
  Interventions: Drug: Fruquintinib and Everolimus

INTERVENTIONS:
Drug: Fruquintinib and Everolimus — Fruquintinib and Everolimus

SUMMARY:
This study will assess the efficacy and safety profile of fruquintinib in combination with everolimus as second line therapy of clear cell renal cell carcinoma patients who progressed after immunotherapy and tyrosine kinase inhibitor.

DETAILED DESCRIPTION:
This study will assess the efficacy and safety profile of fruquintinib in combination with everolimus as second line therapy of clear cell renal cell carcinoma patients who progressed after immunotherapy and tyrosine kinase inhibitor. Patients will receive fruquintinib 4mgQd/5mgQd 21days on/7 days off plus everolimus 5mg Qd as the dose escalation phase indicates.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 and ≤75 years of age
2. Able to Sign informed consent form independently.
3. Stage IV clear cell renal cell carcinoma.
4. Subjects must have progressed after IO-TKI therapy.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1.
6. Subjects must have normal organ and marrow function as defined below:

   * Hemoglobin ≥ 9.0 g/dL;Absolute neutrophil count (ANC) ≥ 1,500/mcL; Platelets ≥ 100,000/mcL, independent of transfusions/growth factors within 3 months of treatment start;
   * Serum potassium ≥ 3.5 mmol/L;
   * Serum total bilirubin ≤ 2.0 x upper limit of normal (ULN) (except in subjects with Gilbert's syndrome who have a total bilirubin > 1.5 x ULN, measure direct and indirect bilirubin and if direct bilirubin is ≤ 1.5 x ULN, subject may be eligible);Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 x ULN;Serum albumin ≥ 3.0 g/dL;Serum creatinine < 2.0 x ULN.

Exclusion Criteria:

1. Have received approved systemic anti-tumor therapy within 2 weeks prior to the first administration, including but not limited to:TKI (TKI with a washout period of 2 weeks or 5 half-lives, whichever is shorter), traditional Chinese medicine treatment (Chinese medicine treatment with anti-tumor indications in the instructions, which can be washed out for 1 week before the first administration), cytokine therapy, etc; Has received any one of the drugs in this study for treatment
2. Participated in or participated in another intervention clinical study within 4 weeks prior to the first administration, except for an observational (non intervention) clinical study or being in the survival follow-up stage of an intervention study;
3. Within 60 days prior to the first medication use, significant surgical procedures (such as craniotomy, thoracotomy, or laparotomy, as defined by the researcher) have been performed;
4. Have undergone any surgery or invasive treatment within 4 weeks prior to the first medication use (fistula surgery requires stable fistula formation for 4 weeks, except for renal/bladder puncture fistula, puncture biopsy, and venous catheterization); Or unhealed wounds, ulcers, fractures, or significant surgery expected during the course of this study (note: local treatment for isolated lesions is acceptable for palliative purposes);
5. Received radiation therapy within one week before the first medication; Received curative radiotherapy (including over 25% bone marrow radiotherapy) within the first 4 weeks of screening;
6. Perform close range radiotherapy (such as implanting radiation particles) within 60 days before the first medication;
7. Toxicity caused by previous anti-tumor therapy prior to initial use that has not recovered to the level specified in the American Cancer Society Adverse Event General Terminology (NCI CTCAE) v5.0 ≤ 1 or inclusion criteria;
8. Allergies to fruquintinib, everolimus or other rapamycin analogues (sirolimus etc), or their excipients;
9. Individuals who have developed other malignant tumors within the 5 years prior to enrollment, excluding clinically cured cervical carcinoma in situ/basal cell carcinoma of the skin/squamous cell carcinoma of the skin/ductal carcinoma in situ of the breast, and localized prostate cancer that has undergone radical treatment;
10. Known to have central nervous system (CNS) metastasis and/or spinal cord compression and/or cancerous meningitis, with a history of leptomeningeal carcinoma;
11. The known history of liver diseases with clinical significance, including those with active viral hepatitis (when hepatitis B virus surface antigen (HBsAg) and or hepatitis B virus core antibody (HbcAb) are positive, hepatitis B B virus (HBV) DNA>10000 copies/mL or>2000 IU/mL; Hepatitis C virus (HCV) antibody positive and HCV RNA positive, or other active hepatitis with clinically significant moderate to severe cirrhosis;
12. The patient currently has digestive tract diseases such as active gastric and duodenal ulcers, ulcerative colitis, or active bleeding from unresectable tumors, or other conditions determined by the researcher that may cause gastrointestinal bleeding or perforation; Or those who have a history of gastrointestinal perforation or fistula and have not recovered after surgical treatment;
13. Cardiovascular diseases with significant clinical significance, including but not limited to acute myocardial infarction, severe/unstable angina, or coronary artery bypass grafting surgery within the first 6 months of screening; Congestive heart failure: New York Heart Association (NYHA) grade ≥ 2; Left ventricular ejection fraction (LVEF)<50%;
14. The patient currently has uncontrolled hypertension (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg) even after receiving standardized treatment;
15. The patient currently has any disease or condition that affects drug absorption, or the patient is unable to administer the medication orally;
16. Patients with evidence of bleeding tendency or medical history within 2 months prior to the first medication (such as black stools, vomiting blood, hemoptysis, bloody stools, etc.), regardless of severity (excluding hemorrhoid bleeding);
17. Have a history of arterial thrombosis or deep vein thrombosis within 6 months before the first medication; Or have experienced stroke events and/or transient ischemic attacks within 12 months; Except for patients with thrombosis caused by implantable intravenous infusion pumps or catheters, or those with superficial venous thrombosis who have stabilized after regular anticoagulation treatment;
18. During screening, it was found that the tumor invaded large vascular structures, such as pulmonary arteries, superior vena cava, or inferior vena cava, and the researcher determined that there was a significant risk of bleeding;
19. May lead to other acute or chronic diseases or abnormal laboratory test values: increase the risk of research participation or drug administration, or interfere with the interpretation of research results, and classify patients as ineligible to participate in this study based on the researcher's judgment;
20. Pregnant (positive pregnancy test) or lactating female patients;
21. Have a history of interstitial lung disease, non infectious pneumonia, or poorly controlled diseases, including pulmonary fibrosis, acute lung disease, etc;
22. Severe chronic or active infections (including pulmonary tuberculosis infection) that require systemic antibacterial, antifungal, or antiviral treatment within 14 days prior to administration; Patients receiving prophylactic antibiotic treatment (such as for preventing urinary tract infections, chronic obstructive pulmonary disease, or tooth extraction);
23. Received live vaccination within 14 days before administration;
24. Known history of HIV infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-02-21 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
MTD (Maximum Tolerated Dose) | 6 month
  the maximum dose in which the proportion of patients who experience dose limited toxicity (DLT) within 28 days after the first dose level is less than or equal to 1/6. When DLT occurs in patients with a dose level greater than 1/6, a dose level lower than this dose level is considered MTD. The MTD dose group requires at least 6 DLT evaluable patients to be confirmed.
ORR (Objective Response Rate) | 1 year
  Based on the evaluable set of tumor efficacy, it is defined as the sum of the proportions of patients with confirmed complete response (CR) or partial response (PR) as the best overall evaluation per RECIST(Response Evaluation Criteria In Solid Tumors )1.1criteria

SECONDARY OUTCOMES:
PFS (Progression Free Survival) | 1 year
  The time from when the patient starts receiving the study drug until disease progression (according to RECIST 1.1) or death occurs, whichever occurs first
DCR (Decease Control Rate ) | 1 year
  The best overall assessment is the sum of the proportions of patients who have confirmed CR, PR, and disease stability (SD) (according to RECIST 1.1)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, China